CLINICAL TRIAL: NCT05094778
Title: A Single-portal Endoscopic Approach Through Subcutaneous Tunnel for Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Collaborators: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShenzhenPH Zhuang03
Record Dates: First submitted 2021-10-02; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; carpal tunnel release; pain; nerve compression syndromes
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Nerve Compression Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-portal group (Other): The patients in single-portal group were treated with single-portal palm approach
  Interventions: Procedure: a single-portal palm approach

INTERVENTIONS:
Procedure: a single-portal palm approach — a single-portal palm approach that passes superficially to palmar aponeurosis, and cut the full transverse carpal ligament.

SUMMARY:
Traditional endoscopic release directly accesses the carpal tunnel and thus carries a higher risk of nerve irritability, even nerve injury. Based on our anatomical study, the investigators developed a new endoscopic technique through a single-portal palm approach that passes superficially to palmar aponeurosis, and cut the full transverse carpal ligament. The investigators will compared the technique with the standard dual-portal endoscopic technique.

DETAILED DESCRIPTION:
Conduct a multi-center, comparison clinical trial according to clinical Trial Reporting Standards (CONSORT). Patients in the single-portal group were treated with a single-portal palm approach that passes superficially to palmar aponeurosis and cut the full transverse carpal ligament. The comparison group were treated with Chow endoscopic technique. In order to assess efficiency of single-portal palm approach, the investigators will compared the technique with the standard dual-portal endoscopic technique. The study was approved by Shenzhen People's Hospital and informed consent was signed.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of carpal tunnel syndrome based on Evidence for Surgical Treatment issued by the British Society for Surgery of the Hand
* Symptoms of carpal tunnel syndrome had lasted>2 months or inadequate responses to the non-surgical treatments≥3 months
* moderate to severe symptoms.

Exclusion Criteria:

* mild symptoms or prior injuries to the extremity
* bilateral wrists involved, a combined nerve compression, gout, diabetes or chronic renal failure.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
The sensibility of the pulps of thumb, index finger, and middle finger (mm) | 3 years
  static 2-point discrimination (2PD) test is used for testing the sensibility of the pulps of digits. The range of normal value is 3 mm--5 mm, and higher scores mean a worse outcome
Severity of symptoms and functional status | 3 years
  The Levine Questionnaire is regarded as a valuable assessment of severity of symptoms and functional status in carpal tunnel syndrome. It is self-administered and is in two sections. The symptoms severity scale is 11 questions and evaluates symptoms regarding severity, frequency, time and kind. The functional status scale is eight questions and evaluates how the syndrome affects daily life.Each question had five ordinal response categories ranging from 1 (no symptoms) to 5 (very severe symptoms). Responses to individual items were averaged to yield an overall score for each scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yongqing Zhuang, Principal Investigator — Shenzhen People's Hospital

REFERENCES:
- [Result] Shi Q, Bobos P, Lalone EA, Warren L, MacDermid JC. Comparison of the Short-Term and Long-Term Effects of Surgery and Nonsurgical Intervention in Treating Carpal Tunnel Syndrome: A Systematic Review and Meta-Analysis. Hand (N Y). 2020 Jan;15(1):13-22. doi: 10.1177/1558944718787892. Epub 2018 Jul 17. PMID 30015499
- [Derived] Wei R, Chen C, Liu Y, Liu Z, Xiong H, Zhang X, Zhuang Y. Endoscopic Release Superficial Rather Than Deep to the Transverse Carpal Ligament for Carpal Tunnel Syndrome Improves Immediate Postoperative Transient Symptomatic Exacerbation With Fewer Absences From Work. Arthroscopy. 2023 Apr;39(4):963-970.e2. doi: 10.1016/j.arthro.2022.09.013. Epub 2022 Oct 5. PMID 36208712